CLINICAL TRIAL: NCT04497857
Title: Academic-Community EPINET (AC-EPINET): Mitigating Barriers to Care PILOT
Brief Title: Academic-Community EPINET (AC-EPINET)
Acronym: AC-EPINET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: University of Michigan (Other); Ohio State University (Other); Vanderbilt University (Other); Tulane University (Other); University of Rochester (Other); Yale University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alan Breier, Raymond E. Houk Professor of Psychiatry, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: epinet; 5R01MH120588-02 (NIH)
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders; Major Depression With Psychotic Features; Bipolar Disorder With Psychotic Features
Keywords: psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSC-SD (Placebo Comparator): Standard clinic-based CSC model treatment. Treatment will be delivered largely in clinic for 12 months.
  Interventions: Other: Coordinated Specialty Care (CSC)
- CSC-TH (Experimental): Telehealth based CSC model treatment. Treatment will be delivered largely through telehealth for 12 months.
  Interventions: Other: Coordinated Specialty Care (CSC)

INTERVENTIONS:
Other: Coordinated Specialty Care (CSC) — CSC care is an evidenced-based, comprehensive specialty care programs for young people in the initial phases of psychotic disorders

SUMMARY:
The investigators propose to examine the effects of CSC services delivered via TH (CSC-TH) versus the standard clinic-based CSC model (CSC-SD) on engagement and outcomes in a 12-month, randomized trial.

DETAILED DESCRIPTION:
160 subjects will be randomized into a 12 month study, to one of two treatment arms. The investigators will assess four important elements of engagement to determine which are most sensitive to TH treatment and mediates effects on hospitalization rates. The investigators will assess acceptability and satisfaction of CSC-TH compared to CSC-SD, and deliver a training manual for implementing TH in CSC clinics and for use in future research. Although this study has exploratory aims consistent with pilot projects, The investigators have incorporated methodological rigor where possible (randomization, powering for hospitalization rate) in order to achieve the most robust data to assess the main study questions and inform future trials.

ELIGIBILITY:
Inclusion Criteria:

1. Between 16 and 35 years of age
2. Able to give informed consent
3. Willing and able to adhere to the study schedule
4. New intakes enrolled in one of the six clinical programs
5. Non-affective (schizophrenia, schizoaffective, schizophreniform) and affective (major depression with psychotic features, bipolar disorder with psychotic features) psychotic disorders with onsets within 5 years of enrollment.

Exclusion Criteria:

1. Known IQ < 70 based on participant report

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Annualized hospitalization rates | 12 months
  To determine if CSC-TH, as compared to CSC-SD, is associated with superior clinical outcomes by counting the number of hospitalizations in a year

SECONDARY OUTCOMES:
Number of participants hospitalized | 12 months
  Count of the number of participants hospitalized (adjusted for time in treatment)
Time (days) to first hospitalization | 12 months
  Count of the time in days to first hospitalization
Symptom outcomes assessed by the Modified Colorado Symptom Index (MCSI) | 12 months
  The modified Colorado Symptom Index (MCSI) is a 14-item, self-report scale designed to assess frequency of positive mood and cognitive symptoms in psychosis. Items are rated on a 5-point Likert-style scale (Not at all, Once during the month, Several times during the month, Several times a week, at least every day). Each item is scored on a 0-4 scale (not at all = 0; at least every day = 4) and added together to give a score between 0 and 56, with higher scores indicating greater emotional distress.
Symptom outcomes assessed by the COMPASS-10 | 12 months
  The COMPASS10 consists of 10 items selected from the COMPASS scale developed for the RAISE ETP study. The COMPASS-10 is a clinician-rated assessment of symptom severity in psychosis. There are 10 items measuring anxiety, asociality, avolition, depression, disorganization, hallucinations, hostility, suicidal ideation or behavior, suspiciousness and unusual thought content. The items are rated on a Likert scale from 0 to 6 (0 = not present, 1 =very mild, 2 = mild, 3 = moderate 4= moderately severe, 5 = severe, 6= very severe), with higher scores indicating increased severity of symptoms. For each item, assessors provide ratings of symptom severity after sufficient information is obtained through probe questions.
Functioning outcomes assessed by the MIRECC-GAF | 12 months
  The MIRECC GAF ( Mental Illness Research, Education, and Clinical Center Global Assessment of Functioning) is a three scale assessment of symptom severity, occupational/school functioning, and social functioning. It is scored from 0-100, with a lower score representing worse symptoms/functioning and higher scores representing better functioning. This assessment has been found to have high levels of reliability, concurrent, and predictive validity. It is completed by a trained rater and is expected to take 5 minutes to complete, as the information needed to score the participants will be gathered in various aspects of the assessment process.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Breier, Principal Investigator — Indiana University
Locations (6):
- United States (6):
  - Prevention and Recovery Center for Early Psychosis, Indianapolis, Indiana
  - Early Psychosis Intervention Clinic-New Orleans (EPIC-NOLA) - Tulane University, New Orleans, Louisiana
  - Program for Risk Evaluation and Prevention (PREP) - University of Michigan, Ann Arbor, Michigan
  - Strong Ties Young Adults Program- University of Rochester Medical Center, Rochester, New York
  - The Early Psychosis Intervention Center (EPICENTER) at Ohio State, Columbus, Ohio
  - Vanderbilt's Early Psychosis Program - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT04497857/ICF_000.pdf